CLINICAL TRIAL: NCT04863755
Title: Change of Lifestyle in Elderly Patients With Type 2 Diabetes and Systemic Arterial Hypertension: Effects of DASH Diet and Physical Activity on Blood Pressure and Insulin Sensitivity
Brief Title: Change of Lifestyle in Elderly Patients With Type 2 Diabetes and Systemic Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2017-0086
Record Dates: First submitted 2021-04-08; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Diabetes; Hypertension
Keywords: Diabetes; Hypertension; Elderly; DASH; Steps
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DASH diet only (Other): Patients receive a DASH diet and orientation to maintain their physical activity
  Interventions: Behavioral: DASH
- DASH diet with pedometer (Other): Patients receive a DASH diet and orientation to increase their physical activity with a pedometer steps count
  Interventions: Behavioral: DASHPED

INTERVENTIONS:
Behavioral: DASH — Patients receive DASH diet orientation and recommended to maintain their usual physical activity
  Arms: DASH diet only
Behavioral: DASHPED — Patients receive DASH diet orientation and recommended to increase their usual activity with the use of a pedometer
  Arms: DASH diet with pedometer

SUMMARY:
Evaluate the effect of lifestyle modification through the adoption of a DASH diet, with and without physical activity guidance, on blood pressure and insulin sensitivity in elderly patients with type 2 diabetes and hypertension.

DETAILED DESCRIPTION:
Data regarding the effects of physical activity and DASH-type diet on blood pressure control in patients with type 2 diabetes and hypertension are scarce in the literature, whether evaluating these isolated interventions or together. In addition, most studies do not measure BP using ABPM, which has a special importance in the assessment of pressure homeostasis in DM or are short-term studies. Were only two studies have been identified in the literature that evaluated the effect of the DASH diet on patients with type 2 DM; however, in both trials, being elderly was not an inclusion criterion. The first was an Iranian study that demonstrated in 31 non-hypertensive patients a significant reduction in BP after 8 weeks of following a DASH diet. In the second ECR, we demonstrated that in 20 hypertensive type 2 DM patients, all using antihypertensive drugs and with uncontrolled BP, a DASH-type diet for 4 weeks associated with physical activity reduced the systolic BP assessed by ABPM by 12.5 mmHg. However, the adopted design did not allow to separate the effect of diet from the effect of physical activity. On the other hand, the effect of a single session of walking followed by a 24-hour ABPM assessment showed a reduction in BP in hypertensive elderly and non-hypertensive patients, also without DM. So far it is not defined in patients with type 2 DM and hypertension, especially the elderly, whether the DASH diet alone is as beneficial for BP as its association with physical activity, particularly, considering the difficulties of performing exercises in this group of patients. This is valuable information, as it would reinforce the role of diet therapy intervention even if in isolation in this age group. Furthermore, the role of the DASH diet with or without physical activity remains unknown on insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or more
* Diabetes Mellitus
* Hypertension with poor control

Exclusion Criteria:

* Glucocorticoid use
* Unstable angina
* Acute myocardial infarction in the last 6 months
* Heart failure classes III and IV
* history of cirrhosis, alcoholism or use of illicit drugs
* Dementia and malignant disease that compromises survival in 5 years
* Serum creatinine greater than 2, 0mg / dl
* BMI> 40 kg / m²
* Physical disability that prevents the use of a pedometer
* Participating in another research project involving any type of intervention.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Blood Pressure at 4 months | Baseline and 4 months
  24 hours ambulatory blood pressure monitoring (ABPM)

SECONDARY OUTCOMES:
Change from Baseline Insulin Sensitivity at 4 months | Baseline and 4 months
  HOMA index (using serum fasting insulin and glucose)
Change from Baseline Glucose Profile at 4 months | Baseline and 4 months
  Fasting glucose and A1C
Change from Baseline Weight at 4 months anthropometric variables | Baseline and 4 months
  weight in kilograms
Change from Baseline BMI at 4 months | Baseline and 4 months
  BMI in kg/m2
Change from Baseline Skeletal muscle mass at 4 months | Baseline and 4 months
  Skeletal muscle mass in Kilograms
Change from Baseline Body fat mass at 4 months | Baseline and 4 months
  Body fat mass in kilograms
Change from Baseline Percent body Fat at 4 months | Baseline and 4 months
  Percent body Fat (%)
Change from Baseline Total cholesterol at 4 months | Baseline and 4 months
  Total cholesterol in mg/dl
Change from Baseline LDL cholesterol at 4 months | Baseline and 4 months
  LDL cholesterol in mg/dl
Change from Baseline Triglycerides at 4 months | Baseline and 4 months
  Triglycerides in mg/dl
Change from Baseline HDL cholesterol at 4 months | Baseline and 4 months
  HDL cholesterol in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Verçoza Viana, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
after publication